CLINICAL TRIAL: NCT05169138
Title: The Effect Of Lavender Essential Oil And Inhalation And Massage Methods On Birth Pain İn Primiparous Women
Brief Title: The Effect Of Lavender Essential Oil On Birth Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Seda Karatopuk, Assistant Lecturer, Near East University, Turkey
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/1367
Record Dates: First submitted 2021-11-26; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Labor Pain; Aromatherapy
Keywords: Labor Pain; Aromatherapy,; Lavender Essential Oil; Aromatherapy with lavender essential oil
MeSH Terms: conditions — Labor Pain | interventions — Massage; lavender oil; Inhalation

STUDY DESIGN:
Intervention Model Description: The research was planned to define the superiority of inhalation and massage methods applied with lavender oil compared to the control group and each other.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- massage group with lavender essential oil (Placebo Comparator): Pregnant women (n:37) who participated in this group were given an intense massage for at least 10 minutes in each phase during the first phase of labor. Visual Analog Pain Scale and McGill Melzack Pain Questionnaire were applied before and after the application, and the process was completed with a total of 6 measurements.
  Interventions: Other: Aromatherapy application /massage with lavender oil
- group of inhalations with lavender essential oil (Placebo Comparator): Pregnant women (n:44) who participated in this group were administered inhalation with lavender oil at an intensity of at least 10 minutes in each phase during the first phase of labor. Visual Analog Pain Scale and McGill Melzack Pain Questionnaire were applied before and after the application, and the process was completed with a total of 6 measurements.
  Interventions: Other: Aromatherapy application / inhalation with lavender oil
- control group (No Intervention): No application was made to the pregnant women (n:40) who participated in this group in each phase of the first phase of labor. Despite this, the Visual Analog Pain Scale and McGill Melzack Pain Questionnaire, which were applied at the beginning of each phase in order to increase the reliability of the results, were re-evaluated 30 minutes after the measurements, even though there was no application, and the process was completed with a total of 6 measurements.

INTERVENTIONS:
Other: Aromatherapy application /massage with lavender oil — The application was applied to 37 pregnant women in total, and the effect of massage with lavender oil on labor pain was investigated.
  Arms: massage group with lavender essential oil
Other: Aromatherapy application / inhalation with lavender oil — The application was applied to 41 pregnant women in total, and the effect of inhalation with lavender oil on labor pain was investigated.
  Arms: group of inhalations with lavender essential oil

SUMMARY:
The study was planned as a randomized controlled trial to determine the effect of lavender oil applied to primiparous women by inhalation and massage methods on labor pain.

DETAILED DESCRIPTION:
In universe of the research; Pregnant women who applied to Adana Seyhan State Hospital's Marsa Gynecology and Obstetrics Additional Service Building and Obstetrics Service and Delivery Room between the dates of the study, accepted to participate in the study voluntarily and who met the research conditions included. Numbers 1-2 of a 6-sided dice determined by the dice rolling system formed the control group (40 pregnant), numbers 3-4 were lavender oil inhalation group (44 pregnant), and numbers 5-6 were lavender oil massage group (37 pregnant).

The research was carried out in three stages for the experimental groups and control groups. First stage; Informed Voluntary Consent Form and Questionnaire were applied to the pregnant women whose groups were determined by the chosen randomization method. Afterwards, for the experimental groups according to the group; 10-minute training sessions were given on the inhalation method or massage method with aromatic lavender essential oil. In the second stage; Data were recorded by dividing the first phase of labor into 3 phases for each group. Visual Analog Pain Scale and McGill Melzack Pain Questionnaire were applied to the experimental groups 6 times, before and 30 minutes after the application. At this stage, no application was made in the control group, the Visual Analog Pain Scales and McGill Melzack Pain Questionnaire were applied at the beginning of each phase, the same forms were repeated after 30 minutes and the data were recorded 6 times in total. In the third stage; In the postpartum period, the study was completed by applying the Postpartum Period Information Collection Form by face-to-face interviews with the experimental groups and the pregnant women in the control group.

ELIGIBILITY:
INCLUSİON CRİTERİA:

* Single pregnancy
* Primiparous gestational age more than 36 weeks (term)
* Cervical dilatation of at least 3 cm
* Pregnants with 3 uterine contractions in a 10-minute period lasting at least 30 seconds
* Cephalic presentation
* Not receiving analgesics, sedatives or anesthetics during labor,
* Not using induction at birth

EXCLUSİON CRİTERİA:

* Multiparity
* cephalopelvic incompatibility
* third trimester bleeding history
* intrauterine growth retardation
* multiple pregnancy
* breech presentation
* subject's withdrawal from clinical trial
* allergy to aromatic lavender essential oil
* addiction (alcohol, smoking)
* obstetric conditions requiring emergency cesarean section
* infertility history
* previous history of diagnosis of an underlying disease
* induction at birth

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only primiparous women can participate in this study.
Enrollment: 121 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | through study completion, an average of 9 month
  It is used to convert some values that cannot be measured numerically into numeric. Two extreme values of the parameter to be evaluated are written at the two ends of a 10 cm line, and the patient is asked to determine where his/her condition is appropriate on this line by drawing a line, putting a dot or placing any sign. For pain; "I have no pain" is written on one end and "very severe pain" is written on the other end and the patient is asked to mark the current situation on the line. The minimum score from the scale is 0, and the maximum score is 10. According to the scale, the highest pain value is expressed with 10 points, while 0 defines the least pain.
McGill Melzack Pain Questionnaire | through study completion, an average of 9 month
  It is a multidimensional pain assessment tool consisting of four parts. At the entrance of the form, personal information of the patient, medical diagnosis-problem, introductory information to determine the location, characteristics, relationship and severity of pain according to the patient's perception are included.
  In the McGill Melzack pain questionnaire, the lowest score is 0 and the highest score is 112. 0 denotes the least pain level and the least pain-related discomfort, while 112 denotes the most severe pain and the most pain-related discomfort.
Questionnaire | through study completion, an average of 9 month
  It was developed by the researcher as a result of literature review and includes 30 questions in total. It was aimed to collect information about the sociodemographic and obstetric anamnesis of pregnant women through the form.
Postpartum Period Data Collection Form | through study completion, an average of 9 month
  It was developed by the researcher as a result of literature review and includes 21 questions in total. Via the form; It is aimed to collect information on labor, newborn characteristics, postpartum mother and baby interaction, and evaluation of mothers' satisfaction with massage or inhalation methods.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Yarıcı, Study Director — Study Director
Locations (1):
- Near East University / Turkish Republic of Northern Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No